CLINICAL TRIAL: NCT06662617
Title: Comparison of the Effects of M-TAPA and TAP Nerve Block Applications on Postoperative Pain Scores and Analgesia Requirements in Laparoscopic Cholecystectomy
Brief Title: Analgesic Effect of M-TAPA and TAPB on Laparoscopic Cholesistectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Hüseyin Özden, associate professor, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-03/03
Record Dates: First submitted 2024-10-24; First posted 2024-10-29 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Post Operative Pain
Keywords: laparoscopic cholecystectomy; m-tapa; tap
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: There are two models for this study. Modified Perichondral Approach Thoracoabdominal Nerve block (M-TAPA block) group, and Transversus Abdominal Plane Block (TAP block) group
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and the outcomes assessor who performs postoperative pain evaluation will not know the group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group M-TAPA (Active Comparator): Patients had bilateral M-TAPA block with 0.25% bupivacaine (total volume of 40 ml) at the end of the surgery for postoperative pain control.
  Interventions: Other: modified thoracoabdominal nerve block through perichondrial approach
- Group TAP (Active Comparator): Patients had bilateral TAP block with 0.25% bupivacaine (total volume of 40 ml) at the end of the surgery for postoperative pain control.
  Interventions: Other: Transversus Abdominal Plane block

INTERVENTIONS:
Other: modified thoracoabdominal nerve block through perichondrial approach — After the patient fell asleep, surgery was not yet started. Following sterile conditions for bilateral M-TAPA block application, the transducer was inserted on the chondrium in the sagittal plane at the 9-10th rib level. Subsequently, a deep angle was created with the probe for visualization of the underside of the costochondrium. The sonovisible needle tip was placed just below the chondrium and saline (5 ml) was injected for site confirmation. After the confirmation, 20 ml of 0.25% bupivacaine was administered for each group for a total of 40 ml of local anesthetic. Blocks were applied using an 80 mm sonovisible needle with a 6-10 MHz linear probe under the guidance of a portable ultrasound. Same procedure applied to the contralateral side.
  Arms: Group M-TAPA
Other: Transversus Abdominal Plane block — After the patient fell asleep, surgery was not yet started. Following sterile conditions for bilateral TAP block application, USG will be placed transversely on the mid-axillary line between the iliac crest and subcostal planes. Using the In Plane technique, the block needle will be advanced into the fascial plane between the internal oblique and transversus abdominis muscles and the location will be confirmed by administering 5 ml of saline . After the confirmation, 20 ml of 0.25% bupivacaine was administered for each group for a total of 40 ml of local anesthetic. Blocks were applied using an 80 mm sonovisible needle with a 6-10 MHz linear probe under the guidance of a portable ultrasound. Same procedure applied to the contralateral side.
  Arms: Group TAP

SUMMARY:
Cholecystectomy is the most frequently performed abdominal surgery in developed nations, with laparoscopic cholecystectomy being recognized as the gold standard technique for treating gallstones.

The efficacy of TAP block for pain relief has been well-documented following laparoscopic cholecystectomy procedures. Recently, m-TAPA block has emerged as an alternative analgesic technique for abdominal surgeries.

This study aims to evaluate and compare the effectiveness of these two analgesic methods in managing postoperative pain after laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Cholecystectomy is the most commonly performed abdominal surgery in developed countries, with laparoscopic cholecystectomy regarded as the gold standard technique for gallstone treatment.

Postoperative pain following laparoscopic cholecystectomy is influenced by several factors, making it a complex and predominantly visceral pain. These factors include phrenic nerve irritation due to CO2 insufflation, abdominal distension, port site incisions, the effects of gallbladder removal, and individual patient characteristics.

Regional analgesia has gained widespread acceptance from both patients and physicians, becoming a key component of multimodal analgesia techniques. The transversus abdominis plane (TAP) block has proven effective in reducing postoperative pain in surgeries such as hysterectomy, cholecystectomy, cesarean section, and colorectal procedures.

The Ultrasound (US)-guided Modified Thoracoabdominal Nerve Block Through Perichondrial Approach (M-TAPA) involves administering a local anesthetic to the underside of the perichondral surface. This technique provides effective analgesia for the anterior and lateral thoracoabdominal regions.

The purpose of this study is to compare the efficacy of US-guided M-TAPA block with TAP block for postoperative analgesia following cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients older than 18 years of age who underwent elective laparoscopic cholecystectomy under general anesthesia and were American Society of
* Anesthesiologists (ASA) I-II-III according to the ASA risk classification.

Exclusion Criteria:

* Patients who did not give consent,
* patients with coagulopathy,
* patients with signs of infection at the block application site,
* patients using anticoagulants,
* patients with local anesthetic drug allergies,
* patients undergoing open surgery,
* patients with unstable hemodynamics,
* patients who could not cooperate during postoperative pain assessment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
numerical rating scale scores | postoperative 24 hours
  numerical rating scale is used for pain assessment. The scores of the numerical rating scale changes between 0 to 10 points. 10 points mean "the most severe pain that the patient ever had". 0 point means "there is no pain." Higher scores mean worse outcome.

SECONDARY OUTCOMES:
total tramadol consumption | postoperative 24 hours
  postoperative analgesic need

CONTACTS AND LOCATIONS:
Locations (1):
- Medicana Sivas Hospital, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No